CLINICAL TRIAL: NCT05790967
Title: The Effect of Sex Education on the Sexual Response and Attitudes Towards Sexuality of Pregnant Women
Brief Title: The Effect of Sex Education on Sexuality of Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NESLİHAN YILMAZ SEZER (Other)
Responsible Party: Sponsor-Investigator, NESLİHAN YILMAZ SEZER, Faculty of Nursing, Ankara University
Organization: Ankara University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 20/189
Record Dates: First submitted 2023-03-17; First posted 2023-03-30 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Pregnancy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education Group (Experimental)
  Interventions: Other: Sexual Education
- CONTROL (No Intervention)

INTERVENTIONS:
Other: Sexual Education — Women in the experimental group will be given education on sexual life during pregnancy. Before the training, preliminary data will be collected and then the participants will be given two hours of individual and face-to-face training.
  Arms: Education Group

SUMMARY:
Aim: In this study, it is aimed to determine the effect of sexual education given to pregnant women on attitudes towards sexuality and sexual response during pregnancy.

The study will be carried out in two different groups. After the women are evaluated in terms of eligibility criteria for the research, the eligible pregnant women will be informed about the research and written informed consent will be obtained from those who accept. Random distribution of pregnant women to study groups will be made using the Block Randomization method. The following applications will be made to the groups.

Education Group: Women in the experimental group will be given education on sexual life during pregnancy. Before the training, preliminary data will be collected and then the participants will be given two hours of individual and face-to-face training.

At the end of the training, homework will be given to pregnant women to practice at home, including "sharing their sexual feelings and thoughts with their spouse, sharing problems and concerns about sexuality during pregnancy, and using alternative ways other than sexual intercourse. In addition, a "Sexual Life in Pregnancy Information Booklet" will be given, and they will be asked to read the information in the booklet and share it with their spouses. After 4 weeks, the data sheets will be applied again.

Control Group: Patients in the control group of the study will not be subjected to any treatment other than the routine procedure. Data collection forms will be applied to the patients in the control group at the beginning of the study and after 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Primigravida
* Having a singleton pregnancy
* Being between 14 -22 weeks of pregnancy
* Living with their partner

Exclusion Criteria:

* Pregnant woman or her partner has a previous diagnosis of sexual dysfunction
* Having a risky situation where sexual intercourse is prohibited during pregnancy by the physician
* Use of psychiatric drugs
* Pregnant woman or her partner has a previous diagnosis of sexual dysfunction
* Having a risky situation where sexual intercourse is prohibited during pregnancy by the physician
* Use of psychiatric drugs such as antidepressants

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2023-03-27 (Actual); Primary Completion 2023-06-29 (Actual); Study Completion 2023-06-29 (Actual)

PRIMARY OUTCOMES:
Change in sexual response | baseline, four weeks later
  Pregnancy Sexual Response Inventory which evaluates sexual activity and sexuality problems in pregnant women, consists of two parts and a total of 38 items. The total score ranges from 0 to 100, with scores between 0-25 as "Very bad", between 25-50 as "Bad", between 50-75 as "Good" and between 75-100 as "Excellent".
Attitude Scale toward Sexuality during Pregnancy Change: | baseline, four weeks later
  Attitude towards Sexuality in Pregnancy consists of 34 items and 3 sub-dimensions. The increase in the total score obtained from the scale indicates that the attitudes towards sexuality during pregnancy are positive, and the decrease in the total score indicates that the attitudes towards sexuality during pregnancy are negative. In addition, the cut-off point of the scale was determined as 111.5.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University Cebeci Hospital, Ankara, Mamak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No